CLINICAL TRIAL: NCT01335750
Title: A Clinical Comparison of Marketed Lens Care Solutions With Avaira Lens Brand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CV-09-64, Sterling IRB 3576
Record Dates: First submitted 2010-10-07; First posted 2011-04-14 (Estimated); Results first posted 2013-03-05 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Corneal Staining
Keywords: corneal staining

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Multipurpose Solution #1 (Experimental): B&L Renu Fresh Multipurpose Solution
  Interventions: Other: Multipurpose Solution #1; Other: Multipurpose Solution #2; Other: Mutlipurpose Solution #3; Other: Multipurpose Solution #4
- Multipurpose Solution #2 (Experimental): OptiFree Replenish Multipurpose Solution
  Interventions: Other: Multipurpose Solution #1; Other: Multipurpose Solution #2; Other: Mutlipurpose Solution #3; Other: Multipurpose Solution #4
- Multipurpose Solution #3 (Experimental): Ciba ClearCare Multipurpose Solution
  Interventions: Other: Multipurpose Solution #1; Other: Multipurpose Solution #2; Other: Mutlipurpose Solution #3; Other: Multipurpose Solution #4
- Multipurpose Solution #4 (Active Comparator): Saline Solution
  Interventions: Other: Multipurpose Solution #1; Other: Multipurpose Solution #2; Other: Mutlipurpose Solution #3; Other: Multipurpose Solution #4

INTERVENTIONS:
Other: Multipurpose Solution #1 — B&L Renu Fresh Multipurpose Solution
Other: Multipurpose Solution #2 — Optifree Replenish Multipurpose Solution
Other: Mutlipurpose Solution #3 — Ciba ClearCare Multipurpose Solution
Other: Multipurpose Solution #4 — Saline Solution

SUMMARY:
This study is a clinical comparison of the biocompatibility of several multipurpose solutions, Renu Fresh, Optifree Replenish, and ClearCare, and saline as a control solution among adapted hydrogel contact lens wearers wearing Avaira (enfilcon A) contact lenses at one research site.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent and HIPAA document read, signed, and dated.
* Visual acuity correctable to 20/30 (Snellen) or better in each eye at distance with hydrogel or silicone hydrogel contact lenses.
* Successfully wearing hydrogel or silicone hydrogel contact lenses on a daily wear basis for at least two weeks prior to the study.

Exclusion Criteria:

* History of hypersensitivity
* Evidence or history of epithelial herpes simplex keratitis (dendritic keratitis; vaccinia, active or recent varicella, viral disease of the cornea and/or conjunctiva and/or eyelids; bacterial infection of the eye; and/or fungal disease of the eye
* One functional eye or a monofit eye
* Ocular conditions such as active acute blepharitis, conjunctival infections, and iritis
* Type 2 (macropunctate) or greater corneal staining in any region in either eye as observed by slit-lamp at Visit 1 of each study period
* Sum of the type of corneal staining greater than or equal to 4 across entire cornea in either eye as observed by slit-lamp at Visit 1 of each study period
* Conjunctival staining covering greater than or equal to 20% in 2 or more corneal regions in either eye as observed by slit-lamp at Visit 1 of each study period
* Conjunctival injection greater than Grade 2 (moderate-diffuse redness) in either eye as observed by slit-lamp at Visit 1 of each study period
* Abnormal lenticular opacity in the visual axis of the lens in either eye
* Use of concomitant topical Rx or over-the-counter (OTC) ocular medications
* History of seasonal allergies with significant ocular side effects which may have an adverse impact on contact lens wear
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Andrasko, OD, MS, Principal Investigator — Erdey/Searcy Eye Group
Locations (1):
- Erdey/Searcy Eye Group, Columbus, Ohio, United States

REFERENCES:
- See also: Click here for more information about similar studies — http://www.StainingGrid.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Multipurpose Solution: To obtain results of a clinical comparison of several multipurpose contact lens solutions among adapted hydrogel lens users wearing Avaira contact lenses
Period: Overall Study
Arm/Group | Multipurpose Solution
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Multipurpose Solution
Number analyzed (Participants) | 32
Age, Continuous [Mean (Full Range); unit: Years] | 32 [23 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 18

OUTCOME MEASURES:

1. Secondary Outcome: Subjective Comfort
Description: Subjective comfort ratings 0-100 (0=causes pain, 100=excellent comfort)
Time Frame: Visit 1: Baseline; Visit 2: 2 hours, Visit 3: 4 hours
Population: Subjective comfort ratings 0-100 (0=causes pain, 100=excellent comfort)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Multipurpose Solution #4: Saline Multipurpose Solution
Arm/Group | Multipurpose Solution #1 | Multipurpose Solution #2 | Multipurpose Solution #3 | Multipurpose Solution #4
Number analyzed (Participants) | 32 | 32 | 32 | 32
units on a scale
  Baseline | 82.9 (15.0) | 80.3 (14.6) | 84.8 (13.4) | 84.7 (14.0)
  2 Hour Period | 83.2 (13.9) | 81.6 (15.8) | 85.6 (13.9) | 83.7 (14.5)
  4 Hour Period | 80.5 (14.7) | 78.0 (18.7) | 83.4 (16.3) | 85.3 (14.5)

2. Secondary Outcome: Subjective Dryness
Description: Subjective dryness ratings 0-100 (0=extremely dry, 100=extremely moist)
Time Frame: Visit 1: Baseline; Visit 2: 2 hours, Visit 3: 4 hours
Population: Subjective dryness ratings 0-100 (0=extremely dry, 100=extremely moist)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multipurpose Solution #1 | Multipurpose Solution #2 | Multipurpose Solution #3 | Multipurpose Solution #4
Number analyzed (Participants) | 32 | 32 | 32 | 32
units on a scale
  Baseline | 84.9 (14.0) | 81.1 (15.3) | 85.0 (14.4) | 85.1 (13.1)
  2 Hour Period | 82.8 (13.2) | 76.9 (19.4) | 83.0 (15.3) | 81.7 (16.6)
  4 Hour Period | 81.4 (15.3) | 76.2 (20.1) | 81.9 (16.8) | 83.1 (17.4)

3. Primary Outcome: Corneal Staining Severity
Description: Severity of staining was recorded for each region using a scale of 0-none to 4-patch >/=1mm. Analysis of staining was performed by averaging the scores from the five regions for each eye, then identifying the subject's worse eye at each visit. Mean total severity was calcuated from all identified eyes for each visit.
Time Frame: Baseline, 2 Hour Period, 4 Hour Period
Population: Severity of staining was recorded for each region using a scale of 0-none to 4-patch >/=1mm. Analysis of staining was performed by averaging the scores from the five regions for each eye, then identifying the subject's worse eye at each visit. Mean total severity was calcuated from all identified eyes for each visit.
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Mutlipurpose Solution #1: Optifree Replenish Multipurpose Solution
- Multipurpose Solution #2: B&L Renu Fresh Multipurpose Solution
Arm/Group | Mutlipurpose Solution #1 | Multipurpose Solution #2 | Multipurpose Solution #3 | Multipurpose Solution #4
Number analyzed (Participants) | 32 | 32 | 32 | 32
units on a scale
  Baseline | 0.01 [0 to 4] | 0.01 [0 to 4] | 0.02 [0 to 4] | 0.01 [0 to 4]
  2 Hour Period | 0.10 [0 to 4] | 0.76 [0 to 4] | 0.05 [0 to 4] | 0.06 [0 to 4]
  3 Hour Period | 0.06 [0 to 4] | 0.59 [0 to 4] | 0.06 [0 to 4] | 0.06 [0 to 4]

4. Primary Outcome: Corneal Staining Area
Description: Analysis of staining area was performed by averaging the values from the five regions for each eye and then identifying the subject's worse eye at each visit. Mean total area was calculated from all identified eyes for each visit.
Time Frame: Baseline, 2 Hour Period, 4 Hour Period
Population: Analysis of staining area was performed by averaging the values from the five regions for each eye and then identifying the subject's worse eye at each visit. Mean total area was calculated from all identified eyes for each visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Multipurpose Solution #1: Optifree Replenish
Arm/Group | Multipurpose Solution #1 | Multipurpose Solution #2 | Multipurpose Solution #3 | Multipurpose Solution #4
Number analyzed (Participants) | 32 | 32 | 32 | 32
units on a scale
  Baseline | 0.1 (0) | 0.1 (0) | 0.2 (0) | 0.1 (0)
  2 Hour Period | 1.2 (2.1) | 17.1 (13.2) | 0.6 (1.3) | 0.7 (1.3)
  3 Hour Period | 0.9 (1.6) | 10.3 (11.4) | 0.8 (1.4) | 0.8 (1.7)

ADVERSE EVENTS:
Arm/Group | Multipurpose Solution
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No